CLINICAL TRIAL: NCT02229071
Title: Donafenib in Advanced Hepatocellular Carcinoma: A Randomized Phase 1B Study of Safety, Efficacy, and Pharmacokinetics
Brief Title: Safety and Efficacy of Donafenib in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGDH1B
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2015-03

CONDITIONS: HCC
Keywords: Donafenib; HCC; Advanced; inoperable; Phase 1B
MeSH Terms: interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donafenib(200mg) (Experimental): Donafenib 200 mg orally twice daily,each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: Donafenib(200mg)
- Donafenib(300mg) (Active Comparator): Donafenib 300 mg orally twice daily,each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: Donafenib(300mg)

INTERVENTIONS:
Drug: Donafenib(200mg) — Donafenib 200mg,bid,po
  Other Names: A Group
  Arms: Donafenib(200mg)
Drug: Donafenib(300mg) — Donafenib 300mg,bid,po
  Other Names: B Group
  Arms: Donafenib(300mg)

SUMMARY:
This phase IB study of donafenib, an oral multikinase inhibitor that targets Raf kinase and receptor tyrosine kinases, is to assess toxicity,efficacy and pharmacokinetics in patients wiht advanced hepatocellular carcinoma (HCC) .

DETAILED DESCRIPTION:
Eligibility Criteria:

* 18 -70 years old;
* Patients with measurable, histologically proven, inoperable HCC;
* Child-Pugh (CP) score of A;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less.
* Patients received prior systemic treatments for HCC before 4 weeks;
* Patients received operate before 3 months;
* Patients received TACE before 4 weeks;
* Life expectancy at least 3 months;
* Adequate hepatic and renal function;
* Adequate hematologic function (platelet count,≥70×109per liter;hemoglobin ≥8.5 g per deciliter);
* Prothrombin time international normalized ratio≤2; or prothrombin time ≤16 seconds;or APTT≤43s;or TT≤21s.

Exclusion Criteria:

* Patients had prior treatment with sorafenib;
* CNS involvement.

Method:

* open-label,randomized,multiceters study;
* 2 dose cohorts: 200mg bid and 300mg bid;
* Patients with advanced HCC(inoperable) and Child-Pugh (CP) A , randomized,receive continuous donafenib either 200mg bid or 300mg bid in 4 weeks cycles;
* Sample size:106 patients(53 patients in each dose cohort).

Endpoints:

* Safety: toxicities are assessed according to CTCAE 3.0;
* TTP:Tumor response is assessed every two cycles using RECISIT1.1 criteria;
* Donafenib pharmacokinetics is measured in plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* 18 -70 years old
* Patients with measurable, histologically proven, inoperable HCC
* Child-Pugh (CP) score of A
* Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less.
* Patients received prior systemic treatments for HCC before 4 weeks
* Patients received operate before 3 months
* Patients received TACE before 4 weeks
* Life expectancy at least 3 months
* Adequate hepatic and renal function
* Adequate hematologic function (platelet count,≥70×109per liter;hemoglobin ≥8.5 g per deciliter)
* Prothrombin time international normalized ratio≤2; or prothrombin time ≤16 seconds;or APTT≤43s;or TT≤21s.

Exclusion Criteria:

* Patients had prior treatment with sorafenib
* CNS involvement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | 1 years
  Patient visits are scheduled every 4 weeks to monitor safety and drug accountability. Patients were monitored for adverse events by use of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0

SECONDARY OUTCOMES:
Time to progression(TTP) | 1 year
  Patient visits are scheduled every 8 weeks to monitor efficacy.TTP is measured from the date of randomisation until disease progression according to RECIST 1.1.

OTHER OUTCOMES:
Time to symptomatic progression(TTSP) | 1 year
  Symtomatic progression is measured with the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-HP) domain of physical wellbeing and additional concerns at baseline and every 4 weeks.TTSP is measured from the date of randomisation until symptomatic progression.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Bi, Doctor, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital,SCU, Chengdu, Sichuan, China